CLINICAL TRIAL: NCT03202589
Title: The PAGET Survey : Pre-operative Assessment for GEriatric Trauma Patients
Brief Title: Assessment for GEriatric Trauma Patients
Acronym: PAGET
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0209
Record Dates: First submitted 2017-06-20; First posted 2017-06-28 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-10

CONDITIONS: Geriatric
Keywords: Preoperative assessement for geriatric patients; FOCUS Echocardiography; Orthopedic; Surgery; Geriatric

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FOCUS Echocardiography — FOCUS Echocardiography

SUMMARY:
Hip fracture is the second indication of surgical management elderly patients. It remains linked with a one-year mortality of 20%-25% according to diiferent governmental agencies, and the incidence reaches 30% for those over 80 years old.

The factors recognized and found to be most correlated with the survival / mortality ratio of patients are age, sex, intervention time, and prior health status.

The aim of a preoperative clinical evaluation is to estimate the benefit-risk balance of different clinical and technical managements and to prepare the postoperative patient outcome. During the last decade, management of hip fracture has improved mainly due to the different recommendations for a multidisciplinary management of perioperative procedures. However, none of them have yet highlighted FOCUS echocardiography as a "routine" examination of the preoperative evaluation as in most noncardiac surgeries.

The objective of this study is to evaluate the preoperative management of these patients: Clinical and biological evaluation, and to analyze the place that would have the FOCUS preoperative echocardiography in the choice of the anesthesia technique resulting from the patient evaluation.That study in a pre-requisite study to evaluate the incidence of FOCUS echocardiography realized by anesthesiologists in the preoperative period in order to define patient's outcome and anesthetic management.

DETAILED DESCRIPTION:
The question is whether the pre-operative routine preoperative echographic evaluation would allow the correction or optimization of any comorbiditie, and / or lead to the modification of the anesthetic management of the patients. Feasibility studies have recently focused on the issue of ultrasound targeted at the patient's bedside. Thus, echocardiography data may have implications for anesthetic but also surgical management.

With the advent of ultraportable ultrasound machines, the limit to routine preoperative bedside use of the ultrasound tool appears to be resolved. The use of point-of-care ultrasounds has proven useful in the management of critical patients in emergency and intensive care units and is recommended in many countries.

Tthe investigators first want to assess the preoperative assessment of elderly and fragile patients admitted urgently for hip surgery. The investigators are setting up a multicenter observational questionnaire for consecutive patients. An electronic questionnaire is distributed via SurveyMonkey to various university hospitals, general hospitals and private institutions in France. The objective of this study is to evaluate the preoperative management of these patients: Clinical, biological evaluation, and analyze the current daily practice regarding the place of POC ultrasound preoperatively; the second question is to know if the choice of the anesthesia technique results from the patient's assessment.

The investigators hope to have a reliable survey of current practices on a group of 500 consecutive patients and then to determine with greater accuracy the first expected real hypothesis for a future prospective randomized multicenter study evaluating the use and impact of preoperative ultrasound assessment versus a control group for perioperative management, complications and outcome of patients undergoing hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 66 or more
* Undergoing hip surgery
* Emergency surgery

Exclusion Criteria:

* - Age less than 66years;
* Non hip surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Preoperative assessement for geriatric patients
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Realization of an ultrasound | 1 day
  Incidence of FOCUS echography

SECONDARY OUTCOMES:
Impact on patient management | 1 day
  Impact on patient management

CONTACTS AND LOCATIONS:
Overall Officials: xavier CAPDEVILA, Study Chair — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
nc